CLINICAL TRIAL: NCT04124250
Title: When is it Appropriate to Stop? Applied Field Research to Develop an M&E Strategy to
Brief Title: East New Britain Province Monitoring & Evaluation
Acronym: ENBP M&E
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other); Washington University School of Medicine (Other); Papua New Guinea Institute for Medical Research (Unknown); Papua New Guinea ENB Provincial Health Authority (Unknown); Papua New Guinea National Department of Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: STUDY20191141
Record Dates: First submitted 2019-10-07; First posted 2019-10-11 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Lymphatic Filariasis Elimination by Mass Drug Administration; Monitoring and Evaluation of Mass Drug Administration for Lymphatic Filariasis; Acceptability of Mass Drug Administration for Lymphatic Filariasis
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood spots from participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Mass Drug Administration with a single co-administered dose of Ivermectin, DEC and Albendazole performed by Provincial and National Health Departments annually for two years

SUMMARY:
While tremendous progress towards elimination of lymphatic filariasis (LF) has been made in the 20 years since the 1997 Fiftieth World Health Assembly, it is unlikely the goal of eliminating LF as a public health problem by 2020 will be achieved. As of 2016, it was estimated that 856 million people are still living in areas with ongoing transmission of LF and require mass drug administration (MDA) [1]. Of the 52 countries that remain endemic and require MDA, 22 (42%) have not started MDA in all endemic implementation units (IUs) [1]. In addition, several countries have found that, despite completing the required number of treatment rounds, the response to the present MDA regimen has been suboptimal in some IUs, requiring additional rounds of MDA.

DETAILED DESCRIPTION:
Although the current two-drug regimen has been successful in many places, it is clear that augmented treatment regimens, other alternative strategies, or both are needed to accelerate global elimination. Fortunately, recent scientific studies, led by the DOLF project at Washington University in St. Louis, found that a three-drug regimen, using all three of the medicines typically delivered as a standard two-drug regimen to prevent LF (ivermectin + albendazole or diethycarbamazine + albendazole), is dramatically more effective for achieving sustained clearance of microfilariae from infected persons [2]. WHO conducted a rigorous and thorough review process of data from safety and efficacy trials of the triple drug regimen. In November, 2017, WHO endorsed and provided updated treatment guidelines that endorsed the use of IDA as a MDA regimen for LF elimination programs [3]. Following WHO's formal approval and release of the alternative treatment guidelines, in late November Merck & Co. committed to increase its Mectizan donation by 100 million treatments annually to eliminate LF [4], making the IDA regimen financially feasible for countries to adopt.

According to the recently published guidelines, WHO recommends the use of annual IDA in settings where onchocerciasis is not co-endemic with LF in districts have not yet started MDA, in areas that have received fewer than 4 effective rounds of MDA, and in areas where MDA results have been suboptimal. These guidelines call for the current epidemiological criteria (<1% microfilaremia or <2% antigenemia) to be applied to sentinel and spot check sites to determine whether the IU is eligible to proceed with the transmission assessment survey (TAS) and for the TAS to be used to base MDA-stopping decisions [3]. While the TAS has proven to be an effective tool for basing stopping decisions under the standard two-drug regimens, it is unclear whether the target age group (6-7 year olds) and epidemiologic target (<2% antigenemia in areas with W. bancrofti and <2% BmR1 antibodies in areas with Brugia spp. infections) are appropriate when IDA is used. Because IDA will result in an accelerated interruption of transmission and because the effects of this regimen on adult worms are not yet fully understood, it is possible that new target populations, infection indicators, sampling strategies, and/or thresholds will be required to determine when it is safe to stop IDA.

The purpose of this protocol is to describe the operational research (OR) that is necessary to develop a set of recommendations for WHO to consider regarding appropriate monitoring and evaluation (M&E) strategies for countries implementing IDA. Generating the information necessary to establish robust M&E guidelines requires a significant OR effort to ensure that all relevant information is collected, innovative strategies are considered, and that the ultimate recommendations are supported by evidence across multiple countries. It is important to emphasize that the study design described in this protocol is not what would be recommended of all countries implementing IDA. This protocol is for OR purposes only, with the goal that study findings will lead to a simplified M&E framework that is feasible for use by national LF elimination programs.

ELIGIBILITY:
Inclusion Criteria:

* All individuals ages 5 years to 80 years living in selected villages will be eligible to enroll.
* Must live in the villages for at least 12 months

Exclusion Criteria:

* Minors ages 4 and under will not be eligible to enroll.
* Lived in selected village for less than 12 months.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Two distinct age groups will be sampled as part of each assessment: children 5-9 years old and adolescents and adults >10 years. The child and adult surveys will be conducted in the same selected clusters; however, the adult survey will be conducted in a subset of the households (HHs) selected for the child survey because there are likely to be more eligible adults per HH than children.
Sampling Method: Non-Probability Sample
Enrollment: 12930 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
To determine the presence of W. bancrofti microfilariae | 3 years
  Perform blood smears of venous blood collected at night
To determine the presence of W. bancrofti circulating antigen | 3 years
  Fingerstick blood will be collected to assess the presence and semi-quantitative levels of circulating filarial antigen using Alere filarial test strips

SECONDARY OUTCOMES:
To determine the presence and frequency anopheline mosquitos infected with lymphatic filariasis (Xenomonitoring) | 3 years
  Mosquitoes will be collected by light traps or human landing catches, anopheline mosquitoes separated, pooled and DNA extracted and the presence of W. bancrofti DNA assessed by PCR
To determine the knowledge and attitudes about lymphatic filariasis and acceptability of the mass drug program for lymphatic filariasis | 2 years
  Prior to mass drug treatment and following treatment randomly selected individuals will be asked to complete a questionnaire and subset of individuals interviewed

CONTACTS AND LOCATIONS:
Locations (1):
- East New Britain Provincial Health Authority, Kokopo, East New Britain Province, Papua New Guinea

REFERENCES:
- [Result] Fischer PU, King CL, Jacobson JA, Weil GJ. Potential Value of Triple Drug Therapy with Ivermectin, Diethylcarbamazine, and Albendazole (IDA) to Accelerate Elimination of Lymphatic Filariasis and Onchocerciasis in Africa. PLoS Negl Trop Dis. 2017 Jan 5;11(1):e0005163. doi: 10.1371/journal.pntd.0005163. eCollection 2017 Jan. No abstract available. PMID 28056015
- [Result] Irvine MA, Stolk WA, Smith ME, Subramanian S, Singh BK, Weil GJ, Michael E, Hollingsworth TD. Effectiveness of a triple-drug regimen for global elimination of lymphatic filariasis: a modelling study. Lancet Infect Dis. 2017 Apr;17(4):451-458. doi: 10.1016/S1473-3099(16)30467-4. Epub 2016 Dec 22. PMID 28012943
- [Result] Schmaedick MA, Koppel AL, Pilotte N, Torres M, Williams SA, Dobson SL, Lammie PJ, Won KY. Molecular xenomonitoring using mosquitoes to map lymphatic filariasis after mass drug administration in American Samoa. PLoS Negl Trop Dis. 2014 Aug 14;8(8):e3087. doi: 10.1371/journal.pntd.0003087. eCollection 2014 Aug. PMID 25122037
- [Result] Rao RU, Nagodavithana KC, Samarasekera SD, Wijegunawardana AD, Premakumara WD, Perera SN, Settinayake S, Miller JP, Weil GJ. A comprehensive assessment of lymphatic filariasis in Sri Lanka six years after cessation of mass drug administration. PLoS Negl Trop Dis. 2014 Nov 13;8(11):e3281. doi: 10.1371/journal.pntd.0003281. eCollection 2014. PMID 25393404
- [Derived] Bun K, Mode B, Susapu M, Salo J, Bjerum C, Payne M, Tisch D, Sekihara M, Giorgi E, Weil GJ, Fischer PU, Robinson L, Laman M, King CL. Alternative approaches for monitoring and evaluation of lymphatic filariasis following mass drug treatment with ivermectin, diethylcarbamazine and albendazole in East New Britain Province, Papua New Guinea. PLoS Negl Trop Dis. 2025 Jan 27;19(1):e0012128. doi: 10.1371/journal.pntd.0012128. eCollection 2025 Jan. PMID 39869653
- See also: World Health Organization. Alternative mass drug administration regimens to eliminate lymphatic filariasis. 2017; — http://apps.who.int/iris/bitstream/10665/259381/1/9789241550161-eng.pdf?ua=1
- See also: Merck Commemorates 30 Years of MECTIZAN® Donation Program Progress | Merck Newsroom Home — http://www.mrknewsroom.com/news-release/corporate-news/merck-commemorates-30-years-mectizan-donation-program-progress